CLINICAL TRIAL: NCT00094510
Title: The Effect of Gabapentin on Prefrontal GABA Concentration and Emotional Processing in Healthy Humans
Brief Title: Effect of Gabapentin on GABA Concentration and Emotional Processing
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050006; 05-M-0006
Record Dates: First submitted 2004-10-19; First posted 2004-10-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-09-03

CONDITIONS: Healthy
Keywords: Prefrontal GABA; Stress; Emotion Recognition; Differential Reward; Gabapentin; GABA; Prefrontal Cortex; Emotional Processing; Healthy Humans; Healthy Volunteer; HV

SUMMARY:
This study will use magnetic resonance spectroscopy (MRS) and the drug gabapentin to examine the role of the brain chemical gamma-amino-butyric acid (GABA) in regulating emotions in healthy people. Gabapentin, which is used to treat epilepsy, increases GABA concentrations in the brain. MRS, similar to magnetic resonance imaging (MRI), is a diagnostic test that uses a magnetic field and radio waves to produce images of the brain.

Non-smoking, healthy normal volunteers between 18 and 60 years of age may be eligible for this study. Candidates are screened with a medical history and physical examination, psychiatric evaluation, blood and urine tests, and an electrocardiogram (EKG).

At three separate clinic visits, participants are given either gabapentin or a placebo (an inactive look-alike capsule). They take placebo at one visit, 600 mg of gabapentin at another visit, and 1200 mg of gabapentin at another visit. One hour after taking the capsules, the amount of GABA in the brain is measured by MRS. For this procedure, the subject lies on a table that moves into the MRI scanner (a narrow cylinder), wearing earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. The procedure lasts about 45 to 60 minutes, during which the patient is asked to lie still for up to a few minutes at a time.

DETAILED DESCRIPTION:
Gamma-aminobutyric acid (GABA) is a major inhibitory neurotransmitter in the forebrain structures, and the GABAergic system has been found to have roles in attentional and learning processes, recognition of aversive stimuli, and regulation of emotion and behavior. Decreases in GABA have been associated with seizures, anxiety and mood disorders. Enhancement of GABA may result in anticonvulsive, anxiolytic, and mood-stabilizing effects.

The GABA system has been proposed as a target for novel antidepressant and mood-stabilizing treatments. Recent studies suggest a GABAergic dysfunction in mood and anxiety disorders. Specifically, reduced GABA levels have been found in the occipital cortex of patients with major depression and panic disorder; and after therapy with selective serotonin reuptake inhibitors, an increase in occipital GABA concentrations has been observed in depressed patients and healthy volunteers.

Gabapentin (GBP) is a relatively novel drug that has been approved for the treatment of epilepsy. The effects of GBP on brain amino acid neurotransmitters are not completely understood. GBP significantly increases brain GABA levels in humans after one hour of the first oral dose, although it does not seem to directly affect GABA-specific enzymes, GABA receptors, and GABA uptake. In vitro, GBP stimulates the enzyme glutamic acid decarboxylase that is involved in the synthesis of GABA.

To date, studies that have examined the mechanism of action of GABA enhancing compounds using magnetic resonance spectroscopy (MRS) measured GABA exclusively in the occipital cortex due to technical limitations. Not surprisingly, associations between occipital GABA levels and cognitive measures and psychiatric symptom severity have not been found.

Thanks to a novel MRS method developed by GE and implemented by NIH, reliable measurements of prefrontal GABA levels are now available. The current study is designed to estimate prefrontal GABA levels in a placebo-controlled double-blind study of GBP. It is aimed at evaluating the novel MRS method to estimate prefrontal GABA levels. Prefrontal GABA levels will be related to prefrontal functions including facial emotion recognition and response control. GABA MRS after GBP/placebo may be used as challenge paradigm for future studies aimed at elucidating GABAergic dysfunctions in mood and anxiety disorders. 10 healthy medication-free human subjects will be examined by GABA magnetic resonance spectroscopy in a controlled trial using placebo, 600mg, and 1200mg GBP.

Given the potential role of GABA in the physiologic stress response, this protocol includes a pilot study that compares prefrontal GABA levels between shock/threat-of-shock and no-threat conditions in healthy volunteers. This part of the study may contribute to the elucidation of the role of the prefrontal GABAergic system in the processing of acute stress.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Family history of mental illness (mood and anxiety disorders, schizophrenia and other psychotic disorders, substance abuse disorders) will be obtained in all 1st degree relatives using the Family Interview of Genetic Studies.
* Healthy Control Samples: 34 healthy subjects (ages 18-60) without a known personal or family history of psychiatric disorders in first-degree relatives will be selected.

EXCLUSION CRITERIA:

* Pregnant females will be excluded due to the potential risk of magnetic field exposure during pregnancy.
* If any subject appears incapable of providing informed consent, they will be excluded from the study.
* Subjects must not have taken centrally active medication for at least 3 weeks prior to the study.
* Subjects will also be excluded if they have: a) medical or neurological illnesses likely to affect physiology or anatomy, i.e. hypertension, cardiovascular disorders, b) a history of drug (including benzodiazepines [BZD]) or alcohol abuse, c) smokers, d) serious suicidal ideation or behavior, e) lactose intolerance, f) caffeine dependency, g) history of allergic reaction to GBP, and h) general MRI exclusion criteria.
* Subjects must exhibit no or only moderate alcohol use.
* Subjects beyond age 60 are excluded because of slower elimination of GBP in older adults, and the age-related increase in brain structural abnormalities.
* In women, there are additional exclusion criteria: i) current pregnancy (as documented by pregnancy testing at screening or at days of the challenge studies), j) current breast feeding, k) lack of reliable contraception method.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-10-14; Study Completion 2010-09-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Petroff OA. GABA and glutamate in the human brain. Neuroscientist. 2002 Dec;8(6):562-73. doi: 10.1177/1073858402238515. PMID 12467378
- [Background] McDonagh J, Stephen LJ, Dolan FM, Parks S, Dutton GN, Kelly K, Keating D, Sills GJ, Brodie MJ. Peripheral retinal dysfunction in patients taking vigabatrin. Neurology. 2003 Dec 23;61(12):1690-4. doi: 10.1212/01.wnl.0000098938.80082.25. PMID 14694031
- [Background] Petroff OA, Hyder F, Rothman DL, Mattson RH. Effects of gabapentin on brain GABA, homocarnosine, and pyrrolidinone in epilepsy patients. Epilepsia. 2000 Jun;41(6):675-80. doi: 10.1111/j.1528-1157.2000.tb00227.x. PMID 10840398